CLINICAL TRIAL: NCT00347425
Title: A Multicenter, Open-Label, Parallel-Group, Randomized, Flexible Dose Study To Evaluate the Safety and Tolerability of Switching From Existing Atypical Antipsychotics to Bifeprunox in Subjects With Schizophrenia or Schizoaffective Disorder
Brief Title: Switch Study of Existing Atypical Antipsychotics to Bifeprunox
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: H. Lundbeck A/S (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Loretta Stallings, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S154.3.020; 2006-004972-11
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia and Schizoaffective Disorder
Keywords: Switch Study; Schizophrenia; Atypical Antipsychotics
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Olanzapine; Risperidone; Quetiapine Fumarate; ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other)
  Interventions: Drug: Aripiprazole; Drug: Olanzapine; Drug: Risperidone; Drug: Quetiapine; Drug: Ziprasidone
- B (Other)
  Interventions: Drug: Aripiprazole; Drug: Olanzapine; Drug: Risperidone; Drug: Quetiapine; Drug: Ziprasidone

INTERVENTIONS:
Drug: Aripiprazole — Abrupt discontinuation of prior anti-psychotic med after a successful eight-day up titration of bifeprunox
  Arms: A
Drug: Olanzapine — Abrupt discontinuation of prior anti-psychotic med after a successful eight-day up titration of bifeprunox
  Arms: A
Drug: Risperidone — Abrupt discontinuation of prior anti-psychotic med after a successful eight-day up titration of bifeprunox
  Arms: A
Drug: Quetiapine — Abrupt discontinuation of prior anti-psychotic med after a successful eight-day up titration of bifeprunox
  Arms: A
Drug: Ziprasidone — Abrupt discontinuation of prior anti-psychotic med after a successful eight-day up titration of bifeprunox
  Arms: A
Drug: Aripiprazole — Cross-tapering during which prior anti-psychotic med will be tapered off at the same time while bifeprunox is being titrated up within 8 days
  Arms: B
Drug: Olanzapine — Cross-tapering during which prior anti-psychotic med will be tapered off at the same time while bifeprunox is being titrated up within 8 days
  Arms: B
Drug: Risperidone — Cross-tapering during which prior anti-psychotic med will be tapered off at the same time while bifeprunox is being titrated up within 8 days
  Arms: B
Drug: Quetiapine — Cross-tapering during which prior anti-psychotic med will be tapered off at the same time while bifeprunox is being titrated up within 8 days
  Arms: B
Drug: Ziprasidone — Cross-tapering during which prior anti-psychotic med will be tapered off at the same time while bifeprunox is being titrated up within 8 days
  Arms: B

SUMMARY:
The study will evaluate the safety and tolerability of switching subjects with schizophrenia or schizoaffective disorder from their existing antipsychotic medication to Bifeprunox.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18-65 years, meeting DSM-IV TR diagnosis of Schizophrenia or Schizoaffective Disorder for whom a switch is indicated

Exclusion Criteria:

* Acutely psychotic or with a current Axis I primary psychiatric diagnosis other than schizophrenia or schizoaffective disorder based on DSM-IV TR criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Successful switch defined as those who complete the 4 weeks core study with no worsening of 2 successive post baseline assessments on the CGIS, exacerbation of EPS, or cardiovascular risk factors (body weight and fasting triglycerides) from baseline. | 4 weeks

SECONDARY OUTCOMES:
Adverse events | 4 weeks
Adverse events | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (122):
- United States (63):
  - Site 148, Birmingham, Alabama
  - Site 194, Little Rock, Arkansas
  - Site 178, Anaheim, California
  - Site 167, Cerritos, California
  - Site 189, Cerritos, California
  - Site 183, Culver City, California
  - Site 140, Garden Grove, California
  - Site 162, La Palma, California
  - Site 190, Long Beach, California
  - Site 173, Oceanside, California
  - Site 175, Paramount, California
  - Site 136, Pasadena, California
  - Site 184, Sacramento, California
  - Site 152, San Diego, California
  - Site 186, San Diego, California
  - Site 133, Santa Ana, California
  - Site 171, Torrance, California
  - Site 197, Boca Raton, Florida
  - Site 156, Gainesville, Florida
  - Site 188, Hialeah, Florida
  - Site 193, Jacksonville, Florida
  - Site 154, Miami, Florida
  - Site 163, North Miami, Florida
  - Site 168, North Miami, Florida
  - Site 166, Orange City, Florida
  - Site 124, Orlando, Florida
  - Site 187, Tampa, Florida
  - Site 161, Atlanta, Georgia
  - Site 128, Augusta, Georgia
  - Site 122, Decatur, Georgia
  - Site 174, Chicago, Illinois
  - Site 164, Indianapolis, Indiana
  - Site 172, Lake Charles, Louisiana
  - Site 182, Shreveport, Louisiana
  - Site 121, Glen Burnie, Maryland
  - Site 159, Detroit, Michigan
  - Site 153, Minneapolis, Minnesota
  - Site 145, Saint Charles, Missouri
  - Site 130, St Louis, Missouri
  - Site 141, St Louis, Missouri
  - Site 142, Clementon, New Jersey
  - Site 180, Kenilworth, New Jersey
  - Site 129, Albuquerque, New Mexico
  - Site 131, Brooklyn, New York
  - Site 181, Cedarhurst, New York
  - Site 169, Jamaica, New York
  - Site 195, New York, New York
  - Site 147, Staten Island, New York
  - Site 127, Chagrin Falls, Ohio
  - Site 176, Cincinnati, Ohio
  - Site 191, Oklahoma City, Oklahoma
  - Site 146, Philadelphia, Pennsylvania
  - Site 179, Philadelphia, Pennsylvania
  - Site 196, Sioux Falls, South Dakota
  - Site 134, Memphis, Tennessee
  - Site 170, Memphis, Tennessee
  - Site 177, Austin, Texas
  - Site 185, Conroe, Texas
  - Site 126, Houston, Texas
  - Site 151, San Antonio, Texas
  - Site 138, Richmond, Virginia
  - Site 198, Spokane, Washington
  - Site 165, Huntington, West Virginia
- Argentina (8):
  - Site 302, Buenos Aires
  - Site 305, Buenos Aires
  - Site 306, Córdoba
  - Site 307, La Plata
  - Site 301, Mendoza
  - Site 304, Mendoza
  - Site 308, Mendoza
  - Site 303, Rosario
- Canada (16):
  - Site 116, Chatham, Ontario
  - Site 117, Mississauga, Ontario
  - Site 100, Calgary
  - Site 101, Claresholm
  - Site 110, Halifax
  - Site 111, Hull
  - Site 107, Kelowna
  - Site 109, Kingston
  - Site 115, Markham
  - Site 112, Medicine Hat
  - Site 108, Orléans
  - Site 106, Ottawa
  - Site 104, Prince Albert
  - Site 102, Sherbrooke
  - Site 114, Victoria
  - Site 113, Winnipeg
- Czechia (9):
  - Site 235, Bolonska
  - Site 234, Jablonova
  - Site 216, Litoměřice
  - Site 233, Na Markvartce
  - Site 213, Olomouc
  - Site 214, Pilsen
  - Site 215, Prague
  - Site 217, Prague
  - Site 236, Rejskovo Namesti
- Estonia (3):
  - Site 231, Paldksi Mnt
  - Site 229, Tartu
  - Site 230, Võru
- France (3):
  - Site 202, Clermont-Ferrand
  - Site 203, Dole
  - Site 201, Saint-Cyr-au-Mont-d'Or
- Hungary (9):
  - Site 206, Balassagyarmat
  - Site 204, Budapest
  - Site 205, Budapest
  - Site 208, Budapest
  - Site 211, Budapest
  - Site 207, Debrecen
  - Site 212, Győr
  - Site 209, Gyula
  - Site 210, Pécs
- Latvia (5):
  - Site 219, Balvi
  - Site 221, Jelgava
  - Site 218, Liepāja
  - Site 222, Riga
  - Site 220, Sigulda
- Lithuania (6):
  - Site 225, Kaunas
  - Site 226, Kaunas
  - Site 223, Klaipėda
  - Site 232, Šilutė
  - Site 224, Vilnius
  - Site 228, Vilnius